CLINICAL TRIAL: NCT05870514
Title: Efficacy and Safety of Fospropofol Disodium Versus Propofol for Deep Sedation in Critically Ill Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaobo Yang, MD (Other)
Responsible Party: Sponsor-Investigator, Xiaobo Yang, MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUHICU202304
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Critical Illness
Keywords: Deep sedation; Fospropofol; Propofol; Intensive care unit
MeSH Terms: conditions — Critical Illness | interventions — fospropofol; Injections; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fospropofol disodium for injection (Experimental): Patients in the experimental group received fospropofol disodium for injection at an initial infusion rate of 10 mg/kg/h and adjusted to maintain a Narcotrend index between 13 and 64.
  Interventions: Drug: Fospropofol disodium for injection
- Propofol (Active Comparator): Patients in the active comparator group received propofol at an initial infusion rate of 3 mg/kg/h and adjusted to maintain a Narcotrend index between 13 and 64.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Fospropofol disodium for injection — Patients in the experimental group received fospropofol disodium for injection at an initial infusion rate of 10 mg/kg/h and adjusted to maintain a Narcotrend index between 13 and 64.
  Arms: Fospropofol disodium for injection
Drug: Propofol — Propofol
  Arms: Propofol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fospropofol disodium for injection compared to propofol for deep sedation in mechanically ventilated ICU patients.

DETAILED DESCRIPTION:
This is a randomized, open-label, small sample study using fospropofol disodium and propofol for deep sedation in mechanically ventilated ICU patients. Subjects are randomized to different treatment groups (including 1 for fospropofol disodium and 1 for propofol). Remifentanil is co-administered with fospropofol or propofol. Efficacy and safety profiles of fospropofol disodium and propofol are to be monitoted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years; Expected to require deep sedation ≥8 hours; Requirement for deep sedation (a Narcotrend index between 13 and 64).

Exclusion Criteria:

* Body mass index (BMI) <18 or >30 kg/m2; Contraindicate or allergic to study drugs; Moribund state; Expected to have a general anesthesia within 8 hours; Myasthenia gravis; Acute hepatitis or serious hepatic dysfunction (Child-Pugh class C); Chronic kidney disease with glomerular filtration rate (GFR) < 29 ml/min/1.73m2; Systolic blood pressure less than 90 mm Hg after appropriate intravenous volume replacement and continuous infusions of 2 vasopressors; Acute severe neurological disorder and any other condition interfering with RASS assessment; Pregnancy or lactation; Unstable angina; Acute myocardial infarction; Left ventricular ejection fraction less than 30%; Heart rate less than 50 beats/min; Second- or third-degree heart block in the absence of a pacemaker; Alcohol abuse or drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of time in the target sedation range without rescue sedation | From start of study to 48 hours
  The percentage of time in the target sedation range without rescue sedation

SECONDARY OUTCOMES:
Adverse events | From start of study to 48 hours
  Incidence rate of adverse events
7-day ventilator free time | From start of study to 7 days
  7-day ventilator free time
Success rate of extubation within 7 days | From start of study to 7 days
  Success rate of extubation within 7 days
Length of ICU stay | From start of study to 28 days
  Length of ICU stay
28-day mortality | From start of study to 28 days
  28-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao X, Gao C, Fang X, Ren L, Zhang H, Tang Y, Yuan Y, Qi H, Shu H, Zou X, Yang X, Shang Y. Fospropofol disodium versus Propofol for deep sedation in critically ill patients: a randomized pilot study. BMC Anesthesiol. 2025 Apr 10;25(1):166. doi: 10.1186/s12871-025-03025-x. PMID 40211146